CLINICAL TRIAL: NCT00278915
Title: An Open-label, Non-Comparative Trial to Evaluate the Safety, Efficacy and Pharmacokinetics of Faslodex (Fulvestrant) in Girls With Progressive Precocious Puberty Associated With McCune-Albright Syndrome
Brief Title: Faslodex in McCune-Albright Syndrome
Acronym: FMAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6992C00044; 2005-004893-26 (EudraCT Number)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Puberty, Precocious; McCune-Albright Syndrome
Keywords: Progressive Precocious Puberty; PPP; McCune-Albright Syndrome; MAS
MeSH Terms: conditions — Puberty, Precocious; Fibrous Dysplasia, Polyostotic | interventions — Fulvestrant

ARMS (1):
- Fulvestrant (Experimental): Participants will receive intramuscular injection of fulvestrant 2 mg/kg or 4 mg/kg (First 10 participants will be dosed at 2 mg/kg then increased to 4 mg/kg. All subsequent participants will be dosed at 4 mg/kg) into the buttock or thigh monthly for 12 months or until the participant demonstrates lack of efficacy based upon one or more of the primary endpoints or experiences a serious drug-related toxicity requiring treatment discontinuation.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Participants will receive intramuscular injection of fulvestrant as stated in arm description.
  Other Names: Faslodex; ZD9238

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness and pharmacokinetics of a study drug called Faslodex (fulvestrant) in the treatment of progressive precocious puberty (PPP) (early puberty) in girls with McCune-Albright syndrome (MAS)

ELIGIBILITY:
Inclusion Criteria:

* Females less than or equal to 10 years of age (prior to 11th birthday)
* Diagnosis of MAS
* PPP associated with MAS

Exclusion Criteria:

* Received any prior treatment for PPP associated with MAS with fulvestrant
* Abnormal platelet count or liver function tests
* Bleeding disorders
* Long term anticoagulation therapy
* Known hypersensitivity to any component of the study drug

Ages: 1 Year to 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2006-01-31 (Actual); Primary Completion 2009-12-08 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Faslodex Medical Science Director, MD, Study Director — AstraZeneca
Locations (16):
- United States (7):
  - Research Site, Birmingham, Alabama
  - Research Site, Miami, Florida
  - Research Site, Lexington, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Salt Lake City, Utah
- France (3):
  - Research Site, Bordeaux
  - Research Site, Bron
  - Research Site, Paris
- Germany (2):
  - Research Site, Erlangen
  - Research Site, Osnabrück
- Research Site, Torino, Italy
- Research Site, Moscow, Russia
- United Kingdom (2):
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sims EK, Garnett S, Guzman F, Paris F, Sultan C, Eugster EA; Fulvestrant McCune-Albright study group. Fulvestrant treatment of precocious puberty in girls with McCune-Albright syndrome. Int J Pediatr Endocrinol. 2012 Sep 22;2012(1):26. doi: 10.1186/1687-9856-2012-26. PMID 22999294
- See also: CSR-D6992C00044.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=404&filename=CSR-D6992C00044.pdf
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6992C00044&attachmentIdentifier=c7f1f38d-0976-4974-9fa9-50e2fcb1b0a4&fileName=Clinical_Study_Report_(CSR)_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at study sites located in France, Germany, Italy, Russian Federation, United Kingdom, and the United States of America.
Pre-assignment Details: A total of 30 participants were enrolled in this study.
Groups:
- Fulvestrant: Participants received intramuscular injection of fulvestrant 2 mg/kg or 4 mg/kg (First 10 participants were dosed at 2 mg/kg then increased to 4 mg/kg. All subsequent participants were dosed at 4 mg/kg) into the buttock or thigh monthly for 12 months or until the participant demonstrates lack of efficacy based upon one or more of the primary endpoints or experiences a serious drug-related toxicity requiring treatment discontinuation.
Period: Overall Study
Arm/Group | Fulvestrant
Started | 30
Completed | 29
Not Completed | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: The full-analysis set (FAS) population included participants who received at least 1 dose of study drug.
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.86 (1.846)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 2
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Frequency of Annualized Days of Vaginal Bleeding on Treatment Compared to Baseline
Description: Vaginal bleeding days are defined as the number of days in which vaginal bleeding, (including spotting) occurred. In order to annualize, a 12-month period is defined as 360 days and a 6-month period is defined as 180 days. Frequency of annualized vaginal bleeding days = [(number of vaginal bleeding days)/(total number of days of the time interval under consideration)] multiplied by 360. Change in frequency is equal to the on-treatment frequency minus the baseline frequency. Diary cards will capture days of vaginal bleeding during the 12-month treatment period. Change in the frequency of annualized days of vaginal bleeding during the 12-month treatment period compared to the 6-month baseline period, based on a worst-case scenario calculation (ie, missing diary card days counted as bleeding days) are reported.
Time Frame: Baseline (6 month pre-treatment observation period) through Month 12 treatment period
Population: The full-analysis set (FAS) population included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: Days per year
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Days per year | -3.6 [-42 to 185]

2. Primary Outcome: Percentage of Participants With Baseline Vaginal Bleeding Who Experienced ≥ 50% Reduction in the Number of Vaginal Bleeding Days on Treatment Compared to Baseline
Description: The percentage change in frequency is defined as 100% times the difference (the on-treatment period frequency minus the baseline period frequency), divided by the baseline period frequency. The percentage of participants with baseline vaginal bleeding days who experienced ≥ 50% reduction in the number of vaginal bleeding days during the 12 month treatment period compared to the 6 month baseline period based on a worst-case approach (ie, missing diary card days counted as bleeding days) are reported.
Time Frame: Baseline (6 month pre-treatment observation period) through Month 12 treatment period
Population: The FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants who had bleeding during the 6 month baseline period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 23
Percentage of Participants | 73.9 [51.6 to 89.8]

3. Primary Outcome: Percentage of Participants With Baseline Vaginal Bleeding Who Experienced Cessation of Vaginal Bleeding Over a 6-month Treatment Period
Description: Percentage of participants with baseline vaginal bleeding who experienced cessation of vaginal bleeding days over a 6-month treatment period based on a worst-case approach (ie, missing diary card days counted as bleeding days) are reported.
Time Frame: Baseline (6-month pre-treatment observation period) through Month 12 treatment period
Population: The FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants who had bleeding during the 6-month baseline period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 23
Percentage of Participants | 78.3 [56.3 to 92.5]

4. Primary Outcome: Percentage of Participants With Baseline Vaginal Bleeding Who Experienced Cessation of Vaginal Bleeding Over the Whole 12-month Treatment Period
Description: Percentage of participants with baseline vaginal bleeding who experienced cessation of vaginal bleeding days over a 12-month treatment period based on a worst-case approach (ie, missing diary card days counted as bleeding days) are reported.
Time Frame: Baseline (6 month pre-treatment observation period) through Month 12 treatment period
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 23
Percentage of Participants | 34.8 [16.4 to 57.3]

5. Primary Outcome: Change in Rate of Bone Age (BA) Advancement Over First 6-month Treatment Period Compared to Baseline
Description: Change in rate of BA advancement over first 6-month treatment period compared to baseline (6-month pre-treatment observation period) is reported. Increase in BA is defined as BA (expressed as fractional years) at end of time period minus BA at beginning of time period (unit: years). Rate of increase in BA for a particular time interval is increase in BA during this time interval adjusted (ie, normalized) for the length of this time interval. Rate of BA advancement is change in BA (years) divided by change in chronological age (CA) (years). Change in rate of increase in BA from baseline period to on-treatment period is defined as increase in BA divided by change in CA (in fractional years) between BA radiograph dates. It is calculated as [(BA6 - BA0)/(CA6 - CA0)] - [(BA0 - BA*)/(CA0 - CA*)], where 6, 0, * stand for first Month 6 Visit, Month 0 Visit, and the 6-month retrospective visit, respectively.
Time Frame: Baseline (6-month pre-treatment observation period) through Month 6 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Ratio | -0.83 (1.507)

6. Primary Outcome: Change in Rate of BA Advancement Over Second 6-month Treatment Period Compared to Baseline
Description: Change in rate of BA advancement over second 6-month treatment period compared to baseline (6-month pre-treatment observation period) is reported. Increase in BA is defined as BA (expressed as fractional years) at end of time period minus BA at beginning of time period (unit: years). Rate of increase in BA for a particular time interval is increase in BA during this time interval adjusted (ie, normalized) for the length of this time interval. Rate of BA advancement is change in BA (years) divided by change in CA (years). Change in rate of increase in BA from baseline period to on-treatment period is defined as increase in BA divided by change in CA (in fractional years) between the BA radiograph dates. It is calculated as [(BA6 - BA0)/(CA6 - CA0)] - [(BA0 - BA*)/(CA0 - CA*)], where 6, 0, * stand for second Month 6 Visit, Month 0 Visit, and the 6-month retrospective visit, respectively.
Time Frame: Baseline (6-month pre-treatment observation period) through second Month 6 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Fulvestrant
Number analyzed (Participants) | 29
Ratio | -1.10 (1.383)

7. Primary Outcome: Change in Rate of BA Advancement Over the Whole 12-month Treatment Period Compared to Baseline
Description: Change in rate of BA advancement over whole 12-month treatment period compared to baseline (6-month pre-treatment observation period) is reported. Increase in BA is defined as BA (expressed as fractional years) at end of time period minus BA at beginning of time period (unit: years). Rate of increase in BA for a particular time interval is increase in BA during this time interval adjusted (ie, normalized) for the length of this time interval. Rate of BA advancement is change in BA (years) divided by change in CA (years). Change in rate of increase in BA from baseline period to on-treatment period is defined as increase in BA divided by change in CA (in fractional years) between the BA radiograph dates. It is calculated as [(BA12 - BA0) / (CA12 - CA0)] - [(BA0 - BA*) / (CA0 - CA*)], where 12, 0, * stand for Month 12 Visit, Month 0 Visit, and the 6-month retrospective visit, respectively.
Time Frame: Baseline (6-month pre-treatment observation period) through Month 12 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Ratio | -0.93 (1.343)

8. Primary Outcome: Change in Growth Velocity (Annualized Growth Velocity in cm/Year) Over First 6-month Treatment Period Compared to Baseline
Description: Change in growth velocity (annualized growth velocity in cm/year) from the baseline (pre-treatment period) to first 6-month treatment period is reported. Growth velocity for a particular time period was calculated as the increase in height over that time period divided by the length of that time period (expressed in cm/year). Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Change in growth velocity was calculated as growth velocity on treatment minus change in growth velocity during baseline.
Time Frame: Baseline (6 month pre-treatment observation period) through first 6-month of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
cm/year | -1.7 (4.35)

9. Primary Outcome: Change in Growth Velocity (Annualized Growth Velocity in cm/Year) Over Second 6-month Treatment Period Compared to Baseline
Description: Change in growth velocity (annualized growth velocity in cm/year) from the baseline (pre-treatment period) to second 6-month treatment period is reported. Growth velocity for a particular time period was calculated as the increase in height over that time period divided by the length of that time period (expressed in cm/year). Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Change in growth velocity was calculated as growth velocity on treatment minus change in growth velocity during baseline.
Time Frame: Baseline (6 month pre-treatment observation period) through second 6-month treatment period (ie, through 12-month treatment period)
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
cm/year | -0.8 (4.49)

10. Primary Outcome: Change in Growth Velocity (Annualized Growth Velocity in cm/Year) Over Whole 12-month Treatment Period Compared to Baseline
Description: Change in growth velocity (annualized growth velocity in cm/year) from the baseline (pre-treatment period) to the 12-month treatment period is reported. Growth velocity for a particular time period was calculated as the increase in height over that time period divided by the length of that time period (expressed in cm/year). Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Change in growth velocity was calculated as growth velocity on treatment minus change in growth velocity during baseline.
Time Frame: Baseline (6 month pre-treatment observation period) through Month 12 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
cm/year | -1.4 (3.69)

11. Primary Outcome: Change in Growth Velocity (Z-score) Over the First 6-month Treatment Period Compared to Baseline
Description: Change in growth velocity (Z-score) from baseline period to the first 6 months of treatment period is reported. The Z-score (also known as Standard Deviation Score [SDS]) is defined as [(growth velocity from the previous visit to the current visit minus mean growth velocity) divided by standard deviation (SD)], where the mean and SD are the age- and gender-specific statistics for growth velocity from the National Center for Health Statistics, Fels study and age is the age at the current visit. Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Z-score of 0 represents the population mean for growth velocity. For McCune-Albright Syndrome, Z-score below mean is a better outcome.
Time Frame: Baseline (6 month pre-treatment observation period) through first 6-month treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Unit on a score
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Unit on a score | -1.60 (4.616)

12. Primary Outcome: Change in Growth Velocity (Z-score) Over the Second 6-month Treatment Period Compared to Baseline
Description: Change in growth velocity (Z-score) from baseline period to the second 6 months of treatment period is reported. The Z-score (also known as SDS) is defined as [(growth velocity from the previous visit to the current visit minus mean growth velocity) divided by SD], where the mean and SD are the age- and gender-specific statistics for growth velocity from the National Center for Health Statistics, Fels study and age is the age at the current visit. Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Z-score of 0 represents the population mean for growth velocity. For McCune-Albright Syndrome, Z-score below mean is a better outcome.
Time Frame: Baseline (6 month pre-treatment observation period) through second 6-month treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Unit on a score
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Unit on a score | -0.64 (4.606)

13. Primary Outcome: Change in Growth Velocity (Z-score) Over the Whole 12-month Treatment Period Compared to Baseline
Description: Change in growth velocity (Z-score) from baseline period to 12 months of treatment period is reported. The Z-score (also known as SDS) is defined as [(growth velocity from the previous visit to the current visit minus mean growth velocity) divided by SD)], where the mean and SD are the age- and gender-specific statistics for growth velocity from the National Center for Health Statistics, Fels study and age is the age at the current visit. Baseline growth velocity was calculated from 6-month observational/retrospective period of the study. Z-score of 0 represents the population mean for growth velocity. For McCune-Albright Syndrome, Z-score below mean is a better outcome.
Time Frame: Baseline (6 month pre-treatment observation period) through Month 12 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Unit on a score
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Unit on a score | -1.14 (4.078)

14. Primary Outcome: Change in Uterine Volume From Baseline to Month 6 as Assessed by Ultrasound
Description: Uterine volume was calculated via ultrasound using the formula: 0.5 multiplied by (longitudinal multiplied by anteroposterior multiplied by transverse), if all 3 linear dimensions were recorded. If all 3 linear dimensions were not recorded, uterine volume was not calculated. Change in uterine volume from baseline to Month 6 was calculated as Month 6 volume (by ultrasound) minus screening visit volume (by ultrasound). Baseline (screening visit) is the pre-treatment baseline visit.
Time Frame: Baseline (pre-treatment baseline visit) and Month 6 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants with data at both time points.
Measure: Median (Full Range); unit: Cubic centimeters
Arm/Group | Fulvestrant
Number analyzed (Participants) | 29
Cubic centimeters | -1.10 [-15.10 to 6.04]

15. Primary Outcome: Change in Uterine Volume From Month 6 to Month 12/Final Visit as Assessed by Ultrasound
Description: Uterine volume was calculated via ultrasound using the formula: 0.5 multiplied by (longitudinal multiplied by anteroposterior multiplied by transverse), if all 3 linear dimensions were recorded. If all 3 linear dimensions were not recorded, uterine volume was not calculated. Change in uterine volume from Month 6 to Month 12/final visit was calculated as Month 12/finial visit volume (by ultrasound) minus Month 6 volume (by ultrasound).
Time Frame: At Month 6 and Month 12/final visit treatment period
Population: as for outcome 14
Measure: Median (Full Range); unit: Cubic centimetres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 28
Cubic centimetres | -0.13 [-11.84 to 4.48]

16. Primary Outcome: Change in Uterine Volume From Baseline to Month 12/Final Visit as Assessed by Ultrasound
Description: Uterine volume was calculated via ultrasound using the formula: 0.5 multiplied by (longitudinal multiplied by anteroposterior multiplied by transverse), if all 3 linear dimensions were recorded. If all 3 linear dimensions were not recorded, uterine volume was not calculated. Change in uterine volume from baseline to Month 12/final visit was calculated as End of Study volume (by ultrasound) minus Screening Visit volume (by ultrasound). Baseline (screening visit) is the pre-treatment baseline visit.
Time Frame: Baseline (pre-treatment screening visit) and Month 12 treatment period
Population: as for outcome 14
Measure: Median (Full Range); unit: Cubic centimeters
Arm/Group | Fulvestrant
Number analyzed (Participants) | 27
Cubic centimeters | -2.44 [-10.20 to 6.56]

17. Primary Outcome: Change in Mean Ovarian Volume From Baseline to Month 6 as Assessed by Ultrasound
Description: The mean ovarian volume was the average of both ovaries. Average volume was calculated as 0.5 multiplied by (volume of left ovary plus volume of right ovary) if both volumes were calculated; otherwise, average ovarian volume was considered missing. The volume of each ovary was calculated via ultrasound using the formula: 0.5 multiplied by longitudinal dimension multiplied by anterior-posterior dimension multiplied by transverse dimension. Change in mean ovarian volume from baseline to Month 6 was calculated as Month 6 mean volume minus Screening Visit mean volume. Baseline (screening visit) is the pre-treatment baseline visit.
Time Frame: Baseline (pre-treatment screening visit) and Month 6 of treatment period
Population: as for outcome 14
Measure: Median (Full Range); unit: Cubic centimetres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 25
Cubic centimetres | 0.10 [-27.62 to 7.96]

18. Primary Outcome: Change Mean in Ovarian Volume From Month 6 to Month 12/Final Visit as Assessed by Ultrasound
Description: The mean ovarian volume was the average of both ovaries. Average volume was calculated as 0.5 multiplied by (volume of left ovary plus volume of right ovary) if both volumes were calculated; otherwise, average ovarian volume was considered missing. The volume of each ovary was calculated via ultrasound using the formula: 0.5 multiplied by longitudinal dimension multiplied by anterior-posterior dimension multiplied by transverse dimension. Change in mean ovarian volume from Month 6 to Month 12/final visit was calculated as Month 12/final visit mean volume minus Month 6 mean volume.
Time Frame: At Month 6 and Month 12/final visit treatment period
Population: as for outcome 14
Measure: Median (Full Range); unit: Cubic centimetres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 24
Cubic centimetres | 0.76 [-4.08 to 9.97]

19. Primary Outcome: Change in Mean Ovarian Volume From Baseline to Month 12/Final Visit as Assessed by Ultrasound
Description: The mean ovarian volume was the average of both ovaries. Average ovarian volume was calculated as 0.5 multiplied by (volume of left ovary plus volume of right ovary) if both volumes were calculated; otherwise, average ovarian volume was considered missing. The volume of each ovary was calculated via ultrasound using the formula: 0.5 multiplied by longitudinal dimension multiplied by anterior-posterior dimension multiplied by transverse dimension. Change in mean ovarian volume from baseline to the end of the study was calculated as End of Study mean volume minus Screening Visit mean volume. Baseline (screening visit) is the pre-treatment baseline visit.
Time Frame: Baseline (pre-treatment baseline visit) and Month 12/final visit treatment period
Population: as for outcome 14
Measure: Median (Full Range); unit: Cubic centimetres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 21
Cubic centimetres | 1.01 [-22.25 to 10.36]

20. Primary Outcome: Mean Clearance of Fulvestrant
Description: Mean clearance of fulvestrant is reported.
Time Frame: Post-dose: Weeks 1, 2, 3, and pre-dose: Week 4 of Month 1 for first 6 participants, then pre-dose steady state samples on 2 occasions between Months 6 and 12 with at least 1 month in between wherein first sample drawn at least 30 days following sixth dose
Population: Population pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study drug and have evaluable PK data.
Measure: Mean (Standard Deviation); unit: Litres/hour
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Litres/hour | 38.4 (11.56)

21. Primary Outcome: Mean Volume of Distribution (V1/F) of Fulvestrant
Description: Total apparent volume of distribution (Vss/F) is the total apparent volume in the body into which Fulvestrant distributes at equilibrium. Vss/F = V1/F + V2/F. V1/F is the volume of the first compartment and V2/F is the volume of the second compartment. V1/F of fulvestrant is reported. The measure of variability presented is the inter-individual error.
Time Frame: as for outcome 20
Population: Population PK analysis set included all participants who received at least 1 dose of study drug and have evaluable PK data.
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Litres | 33000 (NA) — The measure of variability presented is the inter-individual error, not the Standard Error. The inter-individual error = 0.492.

22. Primary Outcome: Mean Volume of Distribution (V2/F) of Fulvestrant
Description: Total apparent volume of distribution (Vss/F) is the total apparent volume in the body into which Fulvestrant distributes at equilibrium. Vss/F = V1/F + V2/F. V1/F is the volume of the first compartment and V2/F is the volume of the second compartment. V2/F of fulvestrant is reported. The measure of variability presented is the inter-individual error.
Time Frame: as for outcome 20
Population: as for outcome 21
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Litres | 32700 (NA) — The measure of variability presented is the inter-individual error, not the Standard Error. The inter-individual error = 0.296.

23. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through 68.7 weeks (maximum observed duration)
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Participants
  Any TEAEs | 27
  Any TESAEs | 9

24. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Clinical laboratory parameter analysis included hematology and clinical chemistry.
Time Frame: Day 1 through 68.7 weeks (maximum observed duration)
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Participants
  Anemia | 1
  Vitamin D Deficiency | 1

25. Primary Outcome: Number of Participants With Compliance to Study Treatment
Description: Number of participants with compliance to study treatment are reported. Treatment compliance was ensured at each treatment visit whether each participant received all protocol-defined injections up until the point they either withdrew from the study or completed the main study period. Compliance with study treatment for each participant for the 12-month treatment period was calculated as total number of injections divided by number of visits between first injection (Month 0) and last injection (at Month 11).
Time Frame: Day 1 through Month 12 of treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Participants | 30

26. Primary Outcome: Number of Participants With Withdrawals From Study Treatment Due to TEAE
Description: Number of participants with withdrawals from study treatment due to TEAE are reported.
Time Frame: Day 1 through 68.7 weeks (maximum observed duration)
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Participants | 0

27. Primary Outcome: Hormone Assay: Serum Oestradiol Level
Description: Serum oestradiol level at Month 12 (final visit) is reported.
Time Frame: Month 12 (final visit) of treatment period
Population: he FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants who were evaluable at the specified time point.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Fulvestrant
Number analyzed (Participants) | 26
pmol/L | 25.95 (30.718)

28. Primary Outcome: Hormone Assay: Serum Luteinizing Hormone (LH) Level
Description: Serum LH level collected at Month 12 (final visit) is reported.
Time Frame: Month 12 (final visit) of treatment period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fulvestrant
Number analyzed (Participants) | 28
IU/L | 0.11 (0.042)

29. Primary Outcome: Hormone Assay: Serum Follicle-stimulating Hormone (FSH) Level
Description: Serum FSH level collected at Month 12 (final visit) is reported.
Time Frame: Month 12 (final visit) of treatment period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Fulvestrant
Number analyzed (Participants) | 29
IU/L | 1.13 (1.024)

30. Primary Outcome: Hormone Assay: Serum Testosterone Level
Description: Serum testosterone level at Month 12 (final visit) is reported.
Time Frame: Month 12 (final visit) of treatment period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Fulvestrant
Number analyzed (Participants) | 28
nmol/L | 0.65 (0.273)

31. Secondary Outcome: Change in Tanner Stage of Breast From Baseline to Month 12/Final Visit
Description: Change in Tanner stage (measure of pubertal progression) of breast from baseline to Month 12/last visit is reported. Tanner stage (breast) is a score of range 1-5 where 1 = no development and 5 = adult breast.
Time Frame: From Baseline (Month 0) through Month 12 treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Unit on a scale | 0.0 [-3 to 2]

32. Secondary Outcome: Change in Tanner Stage of Pubic Hair From Baseline to Month 12/Final Visit
Description: Change in Tanner stage (measure of pubertal progression) of pubic hair from baseline to Month 12/final visit is reported. Tanner stage (pubic hair) is a score of range 1-5 where 1 = no development and 5 = adult pubic hair.
Time Frame: From Baseline (Month 0) through Month 12 treatment period
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: Unit on a scale
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Unit on a scale | 0.0 [-2 to 1]

33. Secondary Outcome: Change in Predicted Adult Height (PAH) From Baseline to Month 12/Final Visit
Description: Change in PAH for children over age 6 is reported. Bone age radiographs were collected retrospectively. PAH equals the current height divided by a factor (the fraction of final adult height) based on current bone age (central read) and current bone age relative to chronological age, classified as retarded, average or advanced. Retarded is defined as current bone age (years) < chronological age (years) minus 1; advanced is defined as current bone age (years) > chronological age (years) plus 1; otherwise, bone age is classified as average. The PAH was summarized using the Bayley and Pinneau method.
Time Frame: From Baseline (screening visit) through Month 12 treatment period
Population: The FAS population included participants who received at least 1 dose of study drug. Here, number of participants analyzed denotes those participants who were analyzed for this endpoint.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Fulvestrant
Number analyzed (Participants) | 17
Centimeter | 0.5 (4.10)

34. Secondary Outcome: Percentage of Participants With McCune-Albright Syndrome (MAS) Associated G Protein α-subunit (Gsα) Mutation
Description: The MAS is caused by an activating mutation in the gene coding for the stimulatory subunit of the G protein, Gsα. The altered Gsα causes autonomous activation of G-protein stimulated cyclic adenosine monophosphate (cAMP) formation, which in the gonads, results in episodic uncontrolled sex steroid production and subsequent pubertal development. For participants who provided separate specific informed consent, the percentage of participants with a Gsα mutation at screening was assessed by molecular analysis of peripheral blood.
Time Frame: Baseline (screening)
Population: The FAS population included participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Fulvestrant
Number analyzed (Participants) | 30
Percentage of participants | 23.3

ADVERSE EVENTS:
Time Frame: Day 1 through 68.7 weeks (maximum observed duration)
Description: The FAS population included participants who received at least 1 dose of study drug.
Arm/Group | Fulvestrant
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 9/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant (N=30)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Viral Infection (Infections and infestations) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Neuromyopathy (Nervous system disorders) | 1 (1)
Tic (Psychiatric disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant (N=30)
Pyrexia (General disorders) | 14 (32)
Injection Site Inflammation (General disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Injection Site Pain (General disorders) | 2 (6)
Abdominal Pain (Gastrointestinal disorders) | 8 (21)
Vomiting (Gastrointestinal disorders) | 8 (12)
Diarrhoea (Gastrointestinal disorders) | 5 (7)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (7)
Toothache (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 2 (6)
Headache (Nervous system disorders) | 8 (20)
Lethargy (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Rhinitis (Infections and infestations) | 6 (14)
Bronchitis (Infections and infestations) | 2 (2)
Ear Infection (Infections and infestations) | 3 (5)
Gastroenteritis (Infections and infestations) | 3 (3)
Otitis Media (Infections and infestations) | 2 (8)
Pharyngitis (Infections and infestations) | 2 (3)
Pharyngitis Streptococcal (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (2)
H1N1 Influenza (Infections and infestations) | 2 (4)
Tonsillitis (Infections and infestations) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (8)
Vaginal Infection (Infections and infestations) | 2 (2)
Varicella (Infections and infestations) | 2 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Ear Pain (Ear and labyrinth disorders) | 4 (9)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Decreased Appetite (Metabolism and nutrition disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hot Flush (Vascular disorders) | 2 (2)
Injection Site Reaction (General disorders) | 2 (5)
Nasopharyngitis (Infections and infestations) | 4 (6)

LIMITATIONS AND CAVEATS:
Data for exploration on body weight and race effect on fulvestrant PK is not available due to small sample size. Data for number and size of ovarian cysts at different time-point were too sparse to produce a meaningful summary, hence not reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.